CLINICAL TRIAL: NCT04415970
Title: Understanding Physiology During Float-REST and the Consequential Effects on Subjective and Objective Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1910751767
Record Dates: First submitted 2020-01-17; First posted 2020-06-04 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-04

CONDITIONS: Sleep Quality
Keywords: Sleep; Sensory deprivation tank; Wearable technology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: We aim to assign participants into one of two different sub-study designs:
  1. Group A: Participants will float for 60 minutes, 2 times a week for 8 weeks or use the sleep pod for 60 minutes, 2 times a week for 8 weeks.
  2. Group B: Participants will engage in a crossover design in which they will participate in both float and nap pod, each for two weeks at a time, twice. The order in which these participants engage in the two recovery modalities will be randomly assigned via statistical package R.
  The only difference between Groups A and B is how often/frequent they engage in the two different modalities. Participants in group A will only do float or Metronap - participants in Group B will do both and alternate every two weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flotation Therapy (Experimental): Participants will utilize flotation sensory deprivation tanks.
  Interventions: Other: Flotation therapy sensory deprivation tank
- Sleep Pod (Active Comparator): Participants will utilize sleep pods with partial sensory deprivation (no light and silence).
  Interventions: Other: Sleep Pod

INTERVENTIONS:
Other: Flotation therapy sensory deprivation tank — Participants will float for 60 minutes, 2 times a week for 8 consecutive weeks or alternate with sleep pod every 2 weeks for 8 weeks. All participants will wear a fitness tracker and a sleep monitoring ring worn on the finger for the duration of the study. Each session will be preceded by a short safety questionnaire and an anxiety index. Following each session, the participant will complete the index again. Participants will also complete morning and evening questionnaires and monthly questionnaires on a smartphone.
  Arms: Flotation Therapy
Other: Sleep Pod — Participants will utilize the sleep pod for 60 minutes, 2 times a week for 8 consecutive weeks or alternate with float every 2 weeks for 8 weeks. All participants will wear a fitness tracker and a sleep monitoring ring worn on the finger for the duration of the study. Each session will be preceded by a short anxiety index. Following each session, the participant will complete the index again. Participants will also complete morning and evening questionnaires and monthly questionnaires on a smartphone.
  Arms: Sleep Pod

SUMMARY:
The objective of this research study is to assess how the implementation of various modern strategies for augmented recovery and physiological monitoring via wearable biotechnologies and subjective measurements affect sleep quality, and other indices of recovery from physical activity.

DETAILED DESCRIPTION:
Flotation therapy uses sensory deprivation tanks that consist of a very large warm water enclosure with a high concentration of Epsom salts to create a completely buoyant environment. This, along with a combination of temperature that is kept equal to skin temperature (94 degrees), allows the subject to eliminate the gravitational effects on the body, and along with lack of sound and low to no light (depending on comfort) allows the brain and body to completely relax for augmented physical and mental recovery. To control for potential changes in sleep quality, quantity, and/or stress and anxiety, a control condition utilizing a Metronap nap station to ascertain the effects of standard, horizontal napping with partial sensory deprivation (no light and silence) compared with floating.

To assess whether or not flotation therapy positively influences sleep and perceptual recovery, participants will float for 60 minutes 2 times a week for 8 weeks, use the sleep pod for 60 minutes 2 times a week for 8 weeks, or take part in a cross-over study where the participant will alternate float and sleep pod every 2 weeks for 8 weeks. All participants may wear a fitness tracker and a sleep monitoring ring worn on the finger for the duration of the study. In addition, daily, per session, monthly, and pre/post-study questionnaires will be submitted via a smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older

Exclusion Criteria:

* Do not have any contagious skin infections or diseases
* Do not have a history of seizures
* Do not have a history of being prone to motion sickness
* An episode of loss of consciousness (last 6-months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change in sleep patterns | Daily from baseline through study completion at 8 weeks
  The OURA Rings is a commercially available wearable device that continuously monitors sleep and sleep quality.
Change in self-report measures | Daily from baseline through study completion at 8 weeks
  Short Recovery and Stress Scale (SRSS)-An 8 item inventory that assess subjective measures of physical, mental, and emotional recovery on a 7 point Likert Scale (0=does not apply at all to 6=fully applies). High values in overall recovery indicate feeling physically and mentally recovered. High values in overall stress indicate feeling overloaded and physically tired.
  End of Day Questionnaire (EoD)-Developed at the Rockefeller Neuroscience Institute (RNI) as a modification of the NASA Task Load Index. This questionnaire addresses subjective measures of workload and stressors that were encountered throughout the day.
  Post-Training Rating of Perceived Exertion Questionnaire-An adaption of the Borg Rating of Perceived Exertion scale, commonly referred to as RPE. The questionnaire requires participants to list the specific activity and the subjective measure of exercise intensity. The scale ranges from 6-20 (6=no exertion that is equivalent to rest and 20=maximal exertion).
Change from baseline in self-report measures | At baseline, at 8 weeks
  Big Five Inventory (BFI)-44 item inventory designed to measure the Big Five Factors of personality on a 5-point Likert Scale. Higher scores indicate a higher tendency for that personality trait (1=disagree strongly to 5=agree strongly).
  Emotion Regulation Questionnaire (ERQ)-10-item scale designed to measure tendency to regulate emotions. Each item is answered on a 7-point Likert Scale (1=strongly disagree to 7=strongly agree). Higher scores indicate a higher emotion regulation strategy.
  Five Facet Mindfulness Questionnaire (FFMQ)-39 item inventory assesses the five facets of mindfulness on a 5-point Likert Scale (1=never or very rarely true and 5=very often or always true). Each facet is tallied and the sum total responses are divided by 39 (number of items). Higher scores indicate higher levels of mindfulness.
  State-Trait Anxiety Index (STAI)-20 item inventory assesses state and trait anxiety. Values range from 20 to 80, with higher scores representing more severe anxiety.
Change in monthly self-report measures | At baseline, at 4 weeks, at 8 weeks
  Acute Recovery and Stress Scale (ARSS)- A 32 item inventory that assess subjective measures of physical, mental, and emotional recovery on a 7 point Likert Scale (0=does not apply at all to 6=fully applies). High values in overall recovery indicate feeling physically and mentally recovered. High values in overall stress indicate feeling overloaded and physically tired.
  Pittsburgh Sleep Quality Index (PSQI)- 19 item inventory with 7 subjective components that assess sleep quality over time. Each component is scored from 0 to 3 (0=very good and 3=very bad). The sum of the components is the global score and ranges 0-21 (0=no difficulty and 21=severe difficulties). The higher the global score, the poorer the sleep quality.
Change in per session self-report measures | 2 times a week through study completion at 8 weeks
  State-Trait Anxiety Index (STAI) - Commonly used measure of state and trait anxiety, and done with 20 very brief questions. Values range from 20 to 80, with higher scores representing more severe anxiety. Participants will take the STAI questionnaire before and after each intervention session.

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States